CLINICAL TRIAL: NCT03728439
Title: Analysis of Delayed Onset Muscle Soreness, Functional Performance, Inflammatory and Ergogenic Response of Light Emitting Diodes (LED) Therapy in Rugby Athletes
Brief Title: Effects of Light Emitting Diodes (LED) Therapy in Rugby Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Recovery in rugby athletes
Record Dates: First submitted 2018-10-03; First posted 2018-11-02 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Phototherapy
Keywords: Recovery; Rugby; Phototherapy

STUDY DESIGN:
Intervention Model Description: This is a randomized crossover (crossover) trial. Participants will be randomized to not receive LED (CO) or have the application of LED therapy at three different times: before (Lpré), in the interval (Lin) and after (Lpós) of the Bangsbo and YoyoIR1 performance tests. At 7, 14 and 21 days after the initial tests, the same test and evaluation protocol will be performed. In addition, 48 hours after each test protocol, functional tests, recovery questionnaire and blood collection will be applied for analysis of creatine kinase.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Before (Experimental): LED applications at the beginning, with a dose of 8 J/cm2, will be performed shortly after the blood collections, with a maximum period of 10 minutes, in which the participants of the other groups should remain in rest passive. At the end of these 10 minutes, a 5 minute warm up will be performed and then the tests will be started.
  Interventions: Device: LED before
- Interval (Experimental): The LED therapy applied in the tests interval will be performed after the first block of tests, with a maximum duration of 10 minutes and dose of 8 J/cm2. Then the second block of maximum tests will be performed.
  Interventions: Device: LED interval
- After (Experimental): LED applications at the end will be performed 10 minutes after the second battery of tests, also with 8 J/cm2 and in the same muscles irradiated in the other moments of application.
  Interventions: Device: LED after
- Baseline (No Intervention): On that day, participants will not receive any intervention.

INTERVENTIONS:
Device: LED before — Phototherapy will be applied through LED therapy equipment, with 15 light emitting diodes that produce 8 joules (J) per diode and 120 joules in total. The muscular regions irradiated will be the quadriceps, hamstrings and triceps sural, with two points of application in each muscle group.
  Arms: Before
Device: LED interval — Phototherapy will be applied through LED therapy equipment, with 15 light emitting diodes that produce 8 joules per diode and 120 joules in total. The muscular regions irradiated will be the quadriceps, hamstrings and triceps sural, with two points of application in each muscle group.
  Arms: Interval
Device: LED after — Phototherapy will be applied through LED therapy equipment, with 15 light emitting diodes that produce 8 joules per diode and 120 joules in total. The muscular regions irradiated will be the quadriceps, hamstrings and triceps sural, with two points of application in each muscle group.
  Arms: After

SUMMARY:
Therapy with light emitting diodes (LED) is a good resource to accelerate the recovery of the athlete and reduce muscle damage caused by exercise. Objective: To evaluate the effects of LED therapy applied at different times on late muscle pain (DOMS), functional performance, inflammatory and ergogenic response of rugby athletes. Methodology: Randomized crossover clinical trial, composed of three groups that will receive treatment with LED at three different times. Sample made up of rugby athletes of both sexes, aged between 18 and 35 years. On the first day of the study, there will be an anamnesis, where the participants will answer questions about personal data, history of injuries and training time, right after the participants receive weight, height, heart rate and measured blood pressure, in addition to collecting a blood sample. to standardize the individual's baseline values. After the initial assessment, participants will be randomized to not receive the LED (CO) or receive LED therapy at three different times: before (Lpré), in the interval (Lin) and after (Lpós) the performance tests. Then, the modified Star Trek Balance Test (SEBTm), the Single Jump Test (SGHT) and the Triple Jump Test (THT) will be performed. After that, the Bangsbo Sprint (BST) test will be performed, followed by the Yo-Yo level 1 intermittent recovery test (Yo-Yo IR1). At the end of this test, the subjects will remain at rest for 10 minutes and will be subjected to the same tests (BST and Yo-Yo IR1) again. They will be measured at the end of the second battery of tests, heart rate, blood pressure, subjective perception of effort, muscle pain threshold, blood samples collected and repeated functional tests. After 48 hours of the performance tests, the blood sample will be collected again, the functional tests carried out and they answered a Stress Recovery Questionnaire for Athletes (RESTQ-Sport-76). At 7, 14 and 21 days after the initial tests, the same test and evaluation protocol will be performed, but the participants will receive LED therapy before, during or after the performance tests, according to their randomization. LED therapy will be performed on the rectus femoris, vastus lateralis and vastus medialis muscles; bilateral femoral, semitendinosus and gastrocnemius biceps.

DETAILED DESCRIPTION:
Randomized crossover clinical trial, composed of three groups that will receive LED treatment at three different times. Sample made up of rugby athletes of both sexes, aged between 18 and 35 years. On the first day of the study, there will be an anamnesis, in which the participants will answer questions about personal data, history of injuries and training time, right after receiving weight, height, heart rate and blood pressure, in addition to collecting a blood sample. standardize the baseline values of the individual. After the initial assessment, participants will be randomized to not receive the LED (CO) or receive LED therapy at three different times: before (Lpré), in the interval (Lin) and after (Lpós) of the performance tests. Then, the modified Star Trek Balance Test (SEBTm), the Single Jump Test (SGHT) and the Triple Jump Test (THT) will be performed. Soon after, the familiarization protocol with the Bangsbo Sprint test (BST) will begin, with the participants positioned close to the initial marker (photocell) and the signal, they must execute a maximum of 34.2 meters, performing seven repetitions, with twenty-five seconds duration for active recovery between sprints. At the end of the sprints, the participant will rest for 10 minutes and then perform the intermittent Yo-Yo level 1 recovery test (Yo-Yo IR1). At the end of this test, participants remain at rest for 10 minutes and then perform the same tests (BST and Yo-Yo IR1) again. At the end of the second battery of tests, heart rate, blood pressure, perceived exertion, blood sample and functional tests will be measured again. After 48 hours of performance tests, blood samples will be collected and functional tests will be carried out, in addition to all participants answering the Stress Recovery Questionnaire for Athletes (RESTQ-Sport-76), to quantify the recovery and psychophysiological stress during the test and recovery days. At 7, 14 and 21 days after the initial tests, the same test and evaluation protocol will be performed, but the participants will receive LED therapy before, during or after the performance tests, according to their randomization. All participants will receive LED therapy at the three times, only the application sequence will be randomized. LED therapy will be performed at two points on the quadriceps, two on the hamstrings and two on the gastrocnemius bilaterally. At each point, irradiation will be applied for 60 seconds, with a wavelength of 850nm (± 20nm) and an energy density of 8 joules per square centimeter (J/cm2).

ELIGIBILITY:
Inclusion Criteria:

* Individuals practicing rugby;
* Juvenile and adult categories;
* Minimum training of three days per week;
* Without history of musculoskeletal injuries in the lower limbs in the last year;
* Without the use of supplements or medicines.

Exclusion Criteria:

* Injuries that make it impossible to perform the tests.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in creatine kinase | Before, immediately after and after 48 hours.
  Analysis of inflammatory and cellular lesion responses with creatine kinase (IU/L) test.
Bangsbo sprint test | During the performance protocol and fatigue performed once a week for four weeks.
  To quantify the performance of rugby players in the Bangsbo sprint test (seconds).
Yo-Yo Intermittent Recovery Test | During the performance protocol and fatigue performed once a week for four weeks.
  To quantify the performance of rugby players in the Yo-Yo Intermittent Recovery Test (meters).

SECONDARY OUTCOMES:
Functional performance in the Star Excursion Balance Test | Before, immediately after and after 48 hours.
  Measure the distance (centimeters) reached with each lower limb in the Star Excursion Balance Test modified.
Functional performance in Single Hop Test and Triple Hop Test | Before, immediately after and after 48 hours.
  Measure the distance (centimeters) reached with each lower limb in the Single Hop Test and in the Triple Hop Test.
Recovery and psychophysiological stress | 48 hours after performance tests
  Will be applied the questionnaire Recovery-Stress Questionnaire for Athletes translated and validated for Portuguese language with the objective of evaluating recovery and psychophysiological stress. Consists of 19 scales (General Stress, Emotional Stress, Social Stress, Conflicts / Pressure, Fatigue, Lack of Energy, Complaints Somatic, Success, Social Recovery, Physical Recovery, General Welfare, Sleep Quality, Intervals, Emotional Exhaustion, Injuries, Fitness, Self Acceptance, Self-Efficacy and Self-Regulation), with four questions on each scale, totaling 76 questions. The values of the scales are calculated by the mean values of the items, which can vary from 0 to 6. High scores on the scales associated with stress activities reflect intense subjective stress, while high scores on the scales associated with recovery reflect many recovery activities.
Changes in blood lactate | Before, immediately after the second Yoyo IR1 and 10 minutes after the end of this test.
  Analysis of effort intensity during performance tests

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Macedo, Principal Investigator — State University of Londrina
Locations (1):
- University Hospital of the State University of Londrina, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferraresi C, Dos Santos RV, Marques G, Zangrande M, Leonaldo R, Hamblin MR, Bagnato VS, Parizotto NA. Light-emitting diode therapy (LEDT) before matches prevents increase in creatine kinase with a light dose response in volleyball players. Lasers Med Sci. 2015 May;30(4):1281-7. doi: 10.1007/s10103-015-1728-3. Epub 2015 Feb 27. PMID 25722067
- [Background] Leal-Junior EC, Vanin AA, Miranda EF, de Carvalho Pde T, Dal Corso S, Bjordal JM. Effect of phototherapy (low-level laser therapy and light-emitting diode therapy) on exercise performance and markers of exercise recovery: a systematic review with meta-analysis. Lasers Med Sci. 2015 Feb;30(2):925-39. doi: 10.1007/s10103-013-1465-4. Epub 2013 Nov 19. PMID 24249354
- [Background] Borsa PA, Larkin KA, True JM. Does phototherapy enhance skeletal muscle contractile function and postexercise recovery? A systematic review. J Athl Train. 2013 Jan-Feb;48(1):57-67. doi: 10.4085/1062-6050-48.1.12. PMID 23672326
- [Background] Nampo FK, Cavalheri V, Ramos Sde P, Camargo EA. Effect of low-level phototherapy on delayed onset muscle soreness: a systematic review and meta-analysis. Lasers Med Sci. 2016 Jan;31(1):165-77. doi: 10.1007/s10103-015-1832-4. Epub 2015 Nov 12. PMID 26563953
- [Background] Pinto HD, Vanin AA, Miranda EF, Tomazoni SS, Johnson DS, Albuquerque-Pontes GM, Aleixo IO Junior, Grandinetti VD, Casalechi HL, de Carvalho PT, Leal-Junior EC. Photobiomodulation Therapy Improves Performance and Accelerates Recovery of High-Level Rugby Players in Field Test: A Randomized, Crossover, Double-Blind, Placebo-Controlled Clinical Study. J Strength Cond Res. 2016 Dec;30(12):3329-3338. doi: 10.1519/JSC.0000000000001439. PMID 27050245